CLINICAL TRIAL: NCT04612998
Title: Combined Spinal Epidural Anesthesia in Obese Patients Undergoing Cesarean Surgery: A Randomised Comparison of Lateral Decubitus and Sitting Positions
Brief Title: Combined Spinal Epidural Anesthesia in Obese Patients Undergoing Cesarean Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet AKSOY, Assoc. Prof. Dr. Mehmet AKSOY, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B.30.2.ATA.0.01.00/11
Record Dates: First submitted 2020-10-23; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Obesity; Pregnancy Related; Cesarean Section Complications; Spinal Anaesthetic Poisoning of Undetermined Intent; Hypotension
Keywords: Combined spinal epidural anesthesia; obesity; cesarean section; lateral decubitus position; sitting position; hypotension
MeSH Terms: conditions — Obesity; Hypotension | interventions — Sitting Position

STUDY DESIGN:
Intervention Model Description: Comparator group consisted of patients performing CSEA in the left lateral decubitus position. Active control group consisted of patients performing CSEA in the sitting position.
Who Masked: Outcomes Assessor
Masking Description: In the recovery room, Visual analogue scale (VAS, 0 cm= no pain, 10 cm= worst pain) scores for pain severity, anesthesia-related side effects (e.g., nausea, vomiting and headache), sensory block time (from the spinal injection to the recovery of T10 dermatome), and the time requiring supplemental analgesics was recorded by an independent observer blinded to the group assignment at 30 min and 1st and 2nd hours post-operatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator group (Sham Comparator): Comparator group consisted of patients performing CSEA in the left lateral decubitus position.
  Interventions: Other: left lateral decubitus position; Drug: The use of intravenous ephedrine.; Drug: The use of intravenous atropine.; Drug: The use of intravenous metoclopramide
- Active control group (Active Comparator): Active control group consisted of patients performing CSEA in the sitting position.
  Interventions: Other: sitting position; Drug: The use of intravenous ephedrine.; Drug: The use of intravenous atropine.; Drug: The use of intravenous metoclopramide

INTERVENTIONS:
Other: left lateral decubitus position — Comparator group consisted of patients performing CSEA in the left lateral decubitus position.
  Arms: Comparator group
Other: sitting position — Active control group consisted of patients performing CSEA in the sitting position.
  Arms: Active control group
Drug: The use of intravenous ephedrine. — Intravenous ephedrine (6 mg) was used to treat hypotension (a 30% decrease in systolic blood pressure compared to preoperative values) during surgery.
Drug: The use of intravenous atropine. — Intravenous atropine (1 mg) was given in case of bradycardia (the heart rate < 45 beats/minute) during surgery.
Drug: The use of intravenous metoclopramide — When nausea and vomiting were observed, intravenous metoclopramide (10 mg) was administered.

SUMMARY:
This study investigated the maternal and fetal effects during performance of CSEA in the left lateral decubitus and sitting positions in obese pregnant women undergoing elective cesarean section.

DETAILED DESCRIPTION:
The study population comprised 100 pregnant women diagnosed with obese aged between 18-45 years, American society of anesthesiologist I and II with full-term gestation undergoing elective cesarean section under combined spinal - epidural anesthesia (CSEA). Women with psychiatric diseases, preeclampsia, pregnancy-induced hypertension or chronic hypertension, diabetes, multiple pregnancies, fetal anomaly and allergy to study drugs were excluded from the study. Also, patients requiring general anesthesia and patients with an average blood pressure below 90 and heart rate less than 50 were excluded. Before performance of CSEA, two groups were formed by randomization. A computer-generated table of random numbers was used for randomization. The CESA was performed in left lateral position in Group I (n=50) and in sitting position in Group II (n=50).

Premedication was not performed in any patient. Before entering the operating room, 10 mL/kg lactated Ringer's solution was given to all patients via IV cannula over 20 minutes. Standard monitoring was performed in the operating room. Before the operation; patients' age, weight, height, ASA physical status and basal hemodynamic parameters were recorded. The CSEA was planned for all patients. All interventions were performed by an experienced anesthesiologist. Patients were appropriately positioned in accordance with the group in which they were included. Group I (n=50) consisted of patients performing CSEA in the left lateral decubitus position. The patient was laid on her left side, the legs were flexed on the abdomen and the chin on the chest. Group II (n=50) consisted of patients performing CSEA in the sitting position. The patient was seated on the edge of the operating table with his feet hanging down, the feet supported by a chair, a pillow was given on her lap, and the patient clung to the pillow. After the skin was sterilized and local infiltration was performed with 2% lidocaine, 18 gauge Tuohy needle (Set for CSEA, Braun®, Melsungen, Germany) was advanced through the midline L2-3 or L3-4 intervertebral spaces with loss of resistance technique. Intrathecally, a 27-gauge pencil point needle was inserted using the needle-through-needle technique. When free cerebrospinal fluid flow was seen, 1.8 ml 0.5% isobaric bupivacaine (9 mg) was administered over 30 seconds. The epidural catheter was advanced 3 cm into the epidural space following the spinal needle was removed. After the catheter was checked with negative pressure, it was secured in place. At the end of the procedure patients were placed in the supine position for operation and the operating table was tilted 20° to the left. Sensory block level was evaluated via pinprick test and it was recorded bilaterally every two minutes. Surgery was initiated following the sensory block reached at the upper level of T6 dermatome. If signs of analgesia were not observed within the first 20 min following the spinal injection, spinal anesthesia was evaluated as failed. In case of failure, additional 5 ml solution of 2% lidocaine was performed via the epidural catheter (5-min intervals, the total dose of 15 mg) until a T6 level of the sensory block was provided. Motor block level was evaluated with Modified Bromage scale (scale 0 = motor block is not available; scale 1 = The patient can do the full flexion of foot and knee, she is unable to hip flexion; scale 2 = The patient can do the full flexion of foot, she is unable to knee and hip flexion; scale 3 = Total motor block is available). General anaesthesia protocol was applied in case of three unsuccessful attempts to reach to intrathecal space. Oxygen was delivered during surgery. Intravenous ephedrine (6 mg) was used to treat hypotension (a 30% decrease in systolic blood pressure compared to preoperative values) during surgery. Intra-venous atropine (1 mg) was given in case of bradycardia (the heart rate < 45 beats/minute) during surgery. When nausea and vomiting were observed, intravenous metoclopramide (10 mg) was administered. The application time of the CSEA, the time from the spinal injection to the development of sensory blockade up to T6 dermatome, operation time (the time from the start of the surgical incision until the end of surgery), highest sensory block level, anesthetic complications and the number of patients required epidural medication during surgery were recorded. Following drug administration to the intrathecal space, intraoperative hemodynamic changes were recorded every 2 min. After surgery was initiated, hemodynamic changes were recorded in 5-minute intervals until the end of the operation. Side effects such as pruritus and nausea, the number of patients requiring ephedrine, atropine or analgesic were recorded. After delivery, 30 IU oxytocin in 500 mL Ringer's lactate solution was given intravenously. Neonatal Apgar scores obtained at 1 and 5 min after delivery and umbilical artery blood gas values were recorded.

After surgery, patients were followed in the recovery room for 120 min. In the recovery room, Visual analogue scale (VAS, 0 cm= no pain, 10 cm= worst pain) scores for pain severity, anesthesia-related side effects (e.g., nausea, vomiting and headache), sensory block time (from the spinal injection to the recovery of T10 dermatome), and the time requiring supplemental analgesics was recorded by an independent observer blinded to the group assignment at 30 min and 1st and 2nd hours post-operatively. In the case of VAS > 3 in a patient, 5 ml solution of 2% lidocaine was given through the epidural catheter. When the motor block had regressed to the T10 level, patients were sent to the clinics.Sample size was calculated as minimum 40 patients in each group, based on data obtained in previous studies, to detect a minimum difference in the requirement of 10 mg ephedrine between the two groups with a power of 90%, a of 0.05. Accordingly, 50 pregnant women were recruited in each group to compensate for potential dropouts.

Data were expressed as mean values ± standard deviation (SD) or number and percentage values. Whether the data has normal distribution was tested using Kolmogorov-Smirnov test. Comparisons were performed using the Mann-Whitney U-test, when data was not normally distributed. Comparisons were performed using the Independent T test in the presence of normally distributed data. The percentage values were compared using chi-square, P<0.05 was considered significant statistically.

ELIGIBILITY:
Inclusion Criteria:

* obese women with full-term gestation
* aged between 18-45 years
* ASA (American society of anesthesiologist) I and II
* undergoing elective cesarean section with combined spinal-epidural anesthesia

Exclusion Criteria:

* psychiatric diseases
* preeclampsia
* pregnancy-induced hypertension
* chronic hypertension
* diabetes
* multiple pregnancies
* fetal anomaly
* allergy to study drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — obese women with full-term gestation
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
ephedrine requirement | Every two minutes during surgery.
  The change in ephedrine requirement during surgery (mg).

SECONDARY OUTCOMES:
atropine requirement | every two minutes during surgery
  The change in atropine requirement during surgery (mg).
analgesic requirement | every five minutes after surgery.
  The change in analgesic requirement during surgery (mg).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet AKSOY, Principal Investigator — Faculty of Medicine, Ataturk University, Erzurum, Turkey
Locations (1):
- Mehmet AKSOY, Erzurum, string:Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No